CLINICAL TRIAL: NCT04214418
Title: Phase 1/2 Open-label Study of Combination Therapy With the MEK Inhibitor, Cobimetinib, Immune Checkpoint Blockade, Atezolizumab, and the AUTOphagy Inhibitor, Hydroxychloroquine in KRAS-mutated Advanced Malignancies
Brief Title: Study of Combination Therapy With the MEK Inhibitor, Cobimetinib, Immune Checkpoint Blockade, Atezolizumab, and the AUTOphagy Inhibitor, Hydroxychloroquine in KRAS-mutated Advanced Malignancies
Acronym: MEKiAUTO
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Toxicity and Lack of Efficacy
Sponsor: Columbia University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Gulam Manji, Assistant Professor of Medicine Division of Hematology/Oncology, Columbia University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AAAS4165; ML41472 (Other: Genentech)
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — cobimetinib; Hydroxychloroquine; atezolizumab

STUDY DESIGN:
Intervention Model Description: The phase 1 portion of the study will be conducted using the time-to-event continue reassessment method (TITE-CRM) using four dose levels. The phase 2 portion of the study will use the recommended phase 2 dose for three cohorts with KRAS mutation - 1. Pancreatic adenocarcinoma; 2. Colorectal adenocarcinoma; and 3. Histology agnostic adenocarcinoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: Maximum Tolerated Dose (MTD) (Experimental): Subjects will be treated with combination therapy at the designated dose levels:
  Dose 1 - Hydroxychloroquine 600mg twice per day, Cobimetinib 40mg, no Atezolizumab Dose 2 - Hydroxychloroquine 600mg twice per day, Cobimetinib 40mg, Atezolizumab 840mg Dose 3 - Hydroxychloroquine 600mg twice per day, Cobimetinib 60mg, Atezolizumab 840mg
  Interventions: Drug: Cobimetinib; Drug: Hydroxychloroquine; Drug: Atezolizumab
- Phase 2: Cohort 1 (Experimental): Advanced Pancreatic Adenocarcinoma (N = 23-67) subjects will receive study treatment based on the MTD determined from Phase 1
  Interventions: Drug: Cobimetinib; Drug: Hydroxychloroquine; Drug: Atezolizumab
- Phase 2: Cohort 2 (Experimental): Advanced Colorectal Adenocarcinoma (N = 20-34) subjects will receive study treatment based on the MTD determined from Phase 1
  Interventions: Drug: Cobimetinib; Drug: Hydroxychloroquine; Drug: Atezolizumab
- Phase 2: Cohort 3 (Experimental): Histology Agnostic Adenocarcinoma (N = 23-56) subjects will receive study treatment based on the MTD determined from Phase 1
  Interventions: Drug: Cobimetinib; Drug: Hydroxychloroquine; Drug: Atezolizumab

INTERVENTIONS:
Drug: Cobimetinib — (40-60 mg) orally once daily (morning) on days 1-21 of each 28-day selective small molecule inhibitor for MEK1 and MEK2
Drug: Hydroxychloroquine — (600mg) orally twice daily on days 1-28 of each 28-day cycle
Drug: Atezolizumab — 840 mg IV on Days 1 and 15 of each cycle humanized IgG1 monoclonal antibody (MAb)
  Other Names: TECENTRIQ; MPDL3280A

SUMMARY:
This research study is for patients with an advanced cancer that carries a mutation in a gene called KRAS. Genes are parts of our DNA which carry instructions for a cell (the smallest component of an body part). In many cancers, the KRAS gene contains errors (mutations) which allows the tumors to grow. The purpose of this study is to determine if combination treatment with atezolizumab, cobimetinib, and hydroxychloroquine is safe, and if it will decrease the size of the tumor and prolong life in patients whose tumors contain this mutation. Cobimetinib and atezolizumab are both approved by the FDA for use in other cancers, but not in some cancer types being studied in this trial. Hydroxychloroquine is FDA approved to treat malaria and other conditions, but has also not been approved for these cancer types. Preliminary results have shown that this combination of drugs is effective at killing cancer cells and shrinking tumors in several KRAS-mutated cancers in animals.

DETAILED DESCRIPTION:
The overall objective of this study is to investigate the safety and preliminary efficacy of combination therapy with cobimetinib and hydroxychloroquine, with or without atezolizumab in patients with KRAS-mutated advanced malignancies. Given that the pre-clinical and clinical benefit from this combination is from within poorly differentiated endocrine carcinoma (PDAC) animal models and human subjects with PDAC and duodenal cancer, we will include at least 12 of the 18 evaluable subjects from PDAC and/or colorectal malignancies. The phase 2 portion of the study will be amended after preliminary safety and efficacy results from phase 1 and other ongoing clinical trials have been analyzed and a summary incorporated within the protocol as an amendment including a rationale of the cohorts to be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or pathological confirmation of malignancy with a KRAS-activating mutation.
2. Extent of disease Advanced disease for which no curable options are available. Subjects who are not deemed candidates for these curative therapies will be eligible if they meet other criteria.
3. Prior treatments

   * Pancreatic adenocarcinoma Subjects must have progressed on or be intolerant of combination therapy containing either 5-Fluorouracil/Capecitabine- and/or gemcitabine-based therapy. Subjects who experienced disease recurrence while receiving adjuvant chemotherapy or within three months of completing adjuvant chemotherapy are eligible.
   * Colorectal adenocarcinoma Subjects must have progressed on or be intolerant of combination therapy containing 5-Fluorouracil/Capecitabine, and must have received Oxaliplatin and Irinotecan.
   * MSI-H/dMMR or NTRK-fusion positive tumors Subjects must have received prior treatment with approved drugs for tumors harboring these aberrations.
   * Histology agnostic cancers other than pancreatic and colorectal adenocarcinoma (see above; Phase 1 and 2) Subjects must have progressed on or be intolerant of all standard of care therapies that result in a median progression free survival benefit of ≥ 8 weeks, or overall response rate of >5%.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
5. Age ≥18 years
6. Adequate hematological and end-organ function (test results from within 14 days prior to initiation of study treatment):

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L without granulocyte colony-stimulating factor support
   * White blood cell (WBC) count ≥ 2.5 x 109/L
   * Lymphocyte count ≥ 0.5 x 109/L
   * Platelet count ≥ 100 x 109/L without transfusion
   * Hemoglobin (Hgb) > 9.0 g/dL
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN), unless elevated secondary to bilary obstruction from the pancreas mass and amenable to decompression prior to initiation of therapy
   * Serum total bilirubin ≤ 1.5 x ULN, unless in patients with known Gilbert disease (≤ 3 x ULN), or unless elevated secondary to bilary obstruction from the pancreas mass and amenable to decompression prior to administration of investigational therapy
   * Albumin ≥ 3.0g/dL
   * Creatinine within ULN or calculated creatinine clearance (CrCl) >50 mL/min using the Cockcroft-Gault formula
   * International Normalized Ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN except for those who are on stable anticoagulation for at least three months.
7. Measurable disease according to Immune-modified Response Evaluation Criteria in Solid Tumors (IM-RECIST) and tumor accessible for fresh biopsy if ten adequate paired biopsied specimens have not been procured (Phase 1)
8. Negative pregnancy test and agree to effective form of contraception.
9. Birth control agreement Fertile men must agree to use an effective method of birth control during the study and for up to 3 months after the last dose of study drug.
10. Informed consent Participants must be willing and able to provide written informed consent prior to any study-related procedures and to comply with all study requirements.
11. Ability to comply Participants must be able to comply with the study protocol, according to the investigator's judgement.
12. Deep venous thrombosis (DVT) testing Participants must have undergone lower extremity dopplers to rule out DVT within the screening period, and undergo therapeutic anticoagulation if evidence of DVT is identified.
13. Venous thromboembolism (VTE) testing Patients deemed at increased risk of VTE based on primary cancer, which includes pancreatic adenocarcinoma, gastric/gastroesophageal junction adenocarcinoma, or central nervous system (CNS) malignancy, are to undergo prophylaxis anticoagulation with enoxaparin. Subjects who are unable to receive enoxaparin ,but deemed at increased risk of VTE will not be eligible and consultation with the Principal Investigator is required.
14. Anticoagulation treatment Subjects who are stable on full-dose anticoagulation medication for at least 8 weeks are considered eligible. However, subjects who have an increased clot burden on full-dose anticoagulation will be considered eligible only with the approval of the Principal Investigator.

Exclusion Criteria:

1. Prior treatment with investigational therapy. Participants may not have had any treatments with investigational therapy within the 28 days prior to initiation of study treatment.
2. Prior radiation therapy Participants may not have had radiation therapy within 2 weeks prior to initiation of study treatment. Participants may not have had previous radiotherapy to 25% or more of the bone marrow.
3. Prior Therapy Participants may not have had systemic chemotherapy within 14 days or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment.

   In addition, the following prior treatment is not allowed during Phase 1 of the study:
   * Receptor tyrosine kinase inhibitors targeting MAP kinase pathway;
   * Any pharmacological agents inhibiting the autophagy pathway.

   In addition, the following prior treatment is not allowed during Phase 2 of the study:
   * T-cell co-stimulating agents or immune checkpoint blockade therapies
   * Receptor tyrosine kinase inhibitors targeting Mitogen-Activated Protein (MAP) kinase pathway;
   * Any pharmacological agents inhibiting the autophagy pathway.
4. Adverse events from prior anti-cancer therapy Participants may not initiate treatment if they have adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1 or better, with the exception of Grade ≤ 2 peripheral neuropathy or any grade alopecia.
5. Patients currently receiving any other investigational agents
6. Concomitant treatment with other anti-neoplastic agents (hormone therapy acceptable)
7. Uncontrolled pleural effusion, pericardial effusion, or ascites
8. Patients with symptomatic brain metastases Subjects with untreated brain metastasis ≤ 1 cm can be considered eligible if deemed asymptomatic by the investigator upon consultation with the medical monitor, and do not require immediate radiation or steroids. Subjects with brain metastasis that is treated and stable for 1 month may be considered eligible if they are asymptomatic and on stable dose of steroids, or if they do not require steroids following successful local therapy.
9. Uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy.
10. Recent major surgery or significant traumatic injury Participants may not have undergone major surgery or experienced significant traumatic injury within 14 days prior to initiating study treatment, or be recovering from a procedure related to adverse events of ≤ Grade 1.
11. Active or history of autoimmune disease or immune deficiency

    With the following exceptions:
    * Patients with a history of autoimmune-related hypothyroidism who are on stable thyroid-replacement hormone are eligible for the study.
    * Patients with controlled Type 1 diabetes mellitus who are on a stable insulin regimen are eligible for the study.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are eligible for the study provided all of following conditions are met:

      * Rash must cover <10% of body surface area;
      * Disease is well-controlled at baseline and requires only low-potency topical corticosteroids;
      * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
12. History of idiopathic pulmonary fibrosis, interstitial lung disease, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan [history of radiation pneumonitis in the radiation field (fibrosis) is permitted].
13. Positive for HIV at screening or any time prior to screening Patients without prior positive HIV test result will undergo an HIV test at screening, unless not permitted under local regulations.
14. Active Hepatitis B virus (HBV) infection (chronic or acute) Defined as having a positive hepatitis B surface antigen (HBsAg) test at screening. Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody test at screening, are eligible for the study.
15. Active hepatitis C virus (HCV) infection Defined as positive HCV antibody test followed by a positive HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
16. Known clinically significant liver disease
17. Active tuberculosis
18. Severe infection Patients may not have had a severe infection within 4 weeks prior to initiation of study treatment. This includes, but is not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia. However, patients who were admitted for biliary tract infection due to bile duct obstruction at time of diagnosis must have a functioning biliary stent (as evidenced by declining total bilirubin and ≤ 2 x ULN) and resolved infection (defined by normalization of elevated white blood cell count, absence of signs of infection) and completion of an antibiotic course (at least a seven-day course) prior to initiation of therapy.
19. Recent antibiotic treatment Patients may not have been treated with therapeutic oral or intravenous (IV) antibiotics within 2 weeks prior to initiation of study treatment, except for biliary tract infection due to bile duct obstruction from the pancreas mass. Patients receiving prophylactic antibiotics are eligible for the study.
20. Significant cardiovascular disease Patient may not have significant cardiovascular disease within 12 months prior to initiation of study treatment, seizure disorder, uncontrolled hypertension, or unstable arrhythmia or unstable angina within 3 months prior to initiation of study treatment.
21. Left ventricular ejection fraction below institutional lower limit of normal or below 50%, whichever is lower
22. Baseline QTcF ≥ 450 ms (males) or ≥ 470 ms (females)
23. Grade ≥ 3 hemorrhage or bleeding event within 28 days prior to initiation of study treatment
24. Prior autologous stem cell, allogeneic stem cell, or solid organ transplantation
25. History of malignancy Patient may not have a history of malignancy other than PDA within 2 years prior to screening, with the exception of those with a negligible risk of metastasis or death.
26. Recent vaccination Patients may not have been treated with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipate the need for such a vaccine during treatment with atezolizumab or within 5 months after the last dose of atezolizumab.
27. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
28. Known allergy or hypersensitivity to 4-aminoquinoline compounds or any of the study drug excipients
29. Recent immunosuppressive treatment

    Patients may not have been treated with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipate the need for systemic immunosuppressive medication during the course of the study, with the following exceptions:
    * Patients who received mineralocorticoids, corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study if receiving equivalent to < 10mg of prednisone daily.
    * Patients who received a one-time pulse dose of systemic immunosuppressant medication are eligible for the study after approval from the Principal Investigator.
30. Inability to swallow medication or malabsorption condition that would alter the absorption of orally administered medications
31. History of retinal pathology

    Specifically, patients will be excluded from study participation if they currently are known to have any risk factors for retinal vein occlusion (RVO), including:
    * Glaucoma with intraocular pressure ≥ 21 mmHg;
    * Grade ≥ 2 serum cholesterol;
    * Grade ≥ 2 hypertriglyceridemia;
    * Grade ≥ 2 uncontrolled hypertension (patients with a history of hypertension controlled with anti-hypertensive medication to Grade ≤ 1 are eligible).
32. Pregnancy and breastfeeding
33. Other contraindicated conditions (opinion of treating investigator)
34. Concomitant strong CYP3A4 inhibitors and inducers Concomitant treatment is permitted if the medication is not expected to interfere with the evaluation of safety or efficacy of the study drug.
35. Uncontrolled psoriasis, porphyria, proximal myopathy or neuropathy
36. Severe depression Subjects hospitalized for depression within the past 2 years, or who have prior suicidal attempts will be excluded.
37. Glucose-6-phosphate dehydrogenase deficiency
38. History of connective tissue disorders
39. Subjects on greater than once daily dose of antacid therapy
40. Concomitant use of any of the following drugs:

    * Digoxin
    * Pharmacological agents known to prolong QT interval
    * Mefloquine or other agents which may lower the convulsive threshold
    * Antiepileptics
    * Methotrexate
    * Cyclosporine
    * Ampicillin
    * Cimetidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gulam Manji, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Data and/or specimens will be sent to the sponsor coded with the subject's unique identifier; the link between the unique identifier and the subject will be maintained by the research staff at Columbia University Medical Center (CUIMC).
Time Frame: End of study
Access Criteria: Coded data

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 27 that signed a consent form, 12 were screen failures and one withdrew consent before randomization. A total of 14 participants were assigned to a treatment arm.
Groups:
- Phase I - Dose Level 1: Hydroxychloroquine 600 mg twice per day and Cobimetinib 40 mg once per day
- Phase I - Dose Level 2: Hydroxychloroquine 600mg twice per day, Cobimetinib 40mg once per day, Atezolizumab 840mg on days 1 and 15 of each cycle
- Phase 1- Dose Level 3: Hydroxychloroquine 600mg twice per day, Cobimetinib 60mg once per day, Atezolizumab 840mg on days 1 and 15 of each cycle
- Phase 2: Cohort 1: Advanced Pancreatic Adenocarcinoma subjects will receive study treatment based on the MTD determined from Phase 1
- Phase 2: Cohort 2: Advanced Colorectal Adenocarcinoma subjects will receive study treatment based on the MTD determined from Phase 1
- Phase 2: Cohort 3: Histology Agnostic Adenocarcinoma subjects will receive study treatment based on the MTD determined from Phase 1
Period: Overall Study
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase 1- Dose Level 3 | Phase 2: Cohort 1 | Phase 2: Cohort 2 | Phase 2: Cohort 3
Started | 10 | 4 | 0 | 0 | 0 | 0
Completed | 8 | 2 | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Zero analyzed in the at Phase 1, dose level 3 and Phase 2 cohorts as the study terminated early and zero participants were assigned to those arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase 1- Dose Level 3 | Phase 2: Cohort 1 | Phase 2: Cohort 2 | Phase 2: Cohort 3 | Total
Number analyzed (Participants) | 10 | 4 | 0 | 0 | 0 | 0 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  |  |  |  | 0
  Between 18 and 65 years | 7 | 2 |  |  |  |  | 9
  >=65 years | 3 | 2 |  |  |  |  | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 |  |  |  |  | 8
  Male | 4 | 2 |  |  |  |  | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 |  |  |  |  | 1
  Not Hispanic or Latino | 9 | 4 |  |  |  |  | 13
  Unknown or Not Reported | 0 | 0 |  |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 |  |  |  |  | 1
  Asian | 0 | 0 |  |  |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  |  |  | 0
  Black or African American | 0 | 0 |  |  |  |  | 0
  White | 9 | 4 |  |  |  |  | 13
  More than one race | 0 | 0 |  |  |  |  | 0
  Unknown or Not Reported | 0 | 0 |  |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 4 |  |  |  |  | 14

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Estimated Maximum Tolerated Dose (MTD) Hydroxychloroquine (HCQ)
Description: The MTD is defined as the dose combination at which 30% of the patients experience a dose-limiting toxicity (DLT) by the end of Cycle 2
Time Frame: 28 days
Measure: Number; unit: mg
Groups:
- All Participants: All participants to receive HCQ 600 mg twice a day
Arm/Group | All Participants
Number analyzed (Participants) | 14
mg | 600

2. Primary Outcome: Phase 1: Estimated Maximum Tolerated Dose (MTD) Cobimetinib
Description: as for outcome 1
Time Frame: 28 days
Measure: Number; unit: mg
Groups:
- All Participants: All participants to receive either 40 mg or 60 mg of Cobimetinib
Arm/Group | All Participants
Number analyzed (Participants) | 14
mg | 40

3. Secondary Outcome: Phase 1: Number of Participants With Treatment-Emergent Adverse Events
Description: Adverse events (AEs) and serious adverse events (SAEs) that are deemed to be related to treatment
Time Frame: Up to 20 weeks
Population: Zero analyzed in the at Phase 1, dose level 3 and Phase 2 cohorts as the study terminated early and zero participants were assigned to these arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase 1- Dose Level 3 | Phase 2: Cohort 1 | Phase 2: Cohort 2 | Phase 2: Cohort 3
Number analyzed (Participants) | 10 | 4 | 0 | 0 | 0 | 0
Participants | 9 | 4 |  |  |  |

ADVERSE EVENTS:
Time Frame: Up to 20 weeks
Description: Adverse events collected systematically at each visit
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase 1- Dose Level 3 | Phase 2: Cohort 1 | Phase 2: Cohort 2 | Phase 2: Cohort 3
All-Cause Mortality (participants affected / at risk) | 10/10 | 4/4 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/10 | 1/4 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 10/10 | 4/4 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Dose Level 1 (N=10) | Phase I - Dose Level 2 (N=4) | Phase 1- Dose Level 3 (N=0) | Phase 2: Cohort 1 (N=0) | Phase 2: Cohort 2 (N=0) | Phase 2: Cohort 3 (N=0)
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | NA | NA | NA | NA
Gastrointestinal disorders (Gastrointestinal disorders) | 1 | 1 | NA | NA | NA | NA
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA | NA
Multi-organ failure (General disorders) | 1 | 0 | NA | NA | NA | NA
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Stroke (Nervous system disorders) | 1 | 0 | NA | NA | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I - Dose Level 1 (N=10) | Phase I - Dose Level 2 (N=4) | Phase 1- Dose Level 3 (N=0) | Phase 2: Cohort 1 (N=0) | Phase 2: Cohort 2 (N=0) | Phase 2: Cohort 3 (N=0)
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 5 | 2 | NA | NA | NA | NA
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA | NA
Alkaline phosphatase increased (Investigations) | 3 | 1 | NA | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA | NA | NA
Anemia (Blood and lymphatic system disorders) | 3 | 0 | NA | NA | NA | NA
Anorexia (Metabolism and nutrition disorders) | 3 | 0 | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA | NA | NA
Ascites (Gastrointestinal disorders) | 2 | 0 | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 6 | 1 | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 1 | 2 | NA | NA | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | NA | NA | NA | NA
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA | NA | NA
Chills (General disorders) | 1 | 0 | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 2 | 1 | NA | NA | NA | NA
Creatinine Phosphokinase Increased (Investigations) | 2 | 1 | NA | NA | NA | NA
Creatinine increased (Investigations) | 1 | 0 | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA | NA
Diarrhea (Gastrointestinal disorders) | 6 | 0 | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 0 | 1 | NA | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 1 | 0 | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | NA | NA | NA | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | NA | NA | NA | NA
Edema face (General disorders) | 1 | 0 | NA | NA | NA | NA
Edema limbs (General disorders) | 1 | 0 | NA | NA | NA | NA
Ejection fraction decreased (Cardiac disorders) | 1 | 0 | NA | NA | NA | NA
Eye disorders (Eye disorders) | 1 | 0 | NA | NA | NA | NA
Fatigue (General disorders) | 5 | 1 | NA | NA | NA | NA
Fever (General disorders) | 1 | 0 | NA | NA | NA | NA
Flatulence (Gastrointestinal disorders) | 2 | 1 | NA | NA | NA | NA
Gastrointestinal disorders (Gastrointestinal disorders) | 1 | 0 | NA | NA | NA | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA | NA | NA
Headache (Nervous system disorders) | 1 | 0 | NA | NA | NA | NA
Hepatic infection (Infections and infestations) | 1 | 0 | NA | NA | NA | NA
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA | NA | NA
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA | NA
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | NA | NA | NA | NA
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | NA | NA | NA | NA
Hypotension (Vascular disorders) | 1 | 1 | NA | NA | NA | NA
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 1 | 1 | NA | NA | NA | NA
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0 | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA | NA | NA
Myocardial infarction (Cardiac disorders) | 1 | 0 | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 4 | 2 | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 2 | 0 | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 2 | 0 | NA | NA | NA | NA
Pain (General disorders) | 1 | 0 | NA | NA | NA | NA
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA | NA | NA
Platelet count decreased (Investigations) | 2 | 1 | NA | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | NA | NA | NA | NA
Psychiatric disorders (Psychiatric disorders) | 1 | 0 | NA | NA | NA | NA
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 1 | NA | NA | NA | NA
Sepsis (Infections and infestations) | 2 | 0 | NA | NA | NA | NA
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA | NA | NA
Thrush (Infections and infestations) | 1 | 0 | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 1 | 0 | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 1 | 0 | NA | NA | NA | NA
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | NA | NA | NA | NA
Urine discoloration (Renal and urinary disorders) | 1 | 0 | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 7 | 1 | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the complete nor any part of the results of the study carried out under this protocol, nor any of the information provided by the sponsor for the purposes of performing the study, will be published or passed on to any third party without the consent of the study sponsor. Any investigator involved with this study is obligated to provide the sponsor with complete test results and all data derived from the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/18/NCT04214418/Prot_SAP_000.pdf